CLINICAL TRIAL: NCT01213550
Title: Effects Of Chlorhexidine Mouthrinse On Peridontopathogens: A Randomized, Placebo-Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Sema Becerik, Ege
Other Study IDs: 07-DIS-27
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: This Study Evaluated the Effectiveness of Chlorhexidine Mouthrinse on Subgingival Microbiota
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine (Experimental)
  Interventions: Drug: Chlorhexidine gluconate
- Placebo mouthrinse (Placebo Comparator)
  Interventions: Drug: Placebo mouthrinse

INTERVENTIONS:
Drug: Chlorhexidine gluconate
  Arms: Chlorhexidine
Drug: Placebo mouthrinse
  Arms: Placebo mouthrinse

SUMMARY:
The aim of this study is to evaluate the therapeutic effectiveness of chlorhexidine mouthrinse on gingival inflammation and subgingival microbiota in addition to daily mechanical plaque control in a population with established gingivitis.

DETAILED DESCRIPTION:
Failure to perform oral hygiene adequately at the gingival margin results in the formation of a pathogenic plaque that has the potential to initiate gingivitis and in some individuals to progress to periodontitis. However, factors, such as dexterity and motivation, can limit the effectiveness of daily self-performed oral hygiene. The use of a chemical plaque-inhibitory mouthrinse as an adjunct to toothbrushing may improve the oral health of individuals who are inadequate in mechanical plaque control in maintaining gingival health.

Chlorhexidine (CHX) has been effectively used in the treatment of gingival inflammation and can be considered as the gold standard for oral antiseptics.

The effectiveness of CHX in reducing the formation of dental plaque and preventing gingivitis in addition to professional mechanical debridement were studied in several clinical studies, but there is limited number of studies investigating the effects of CHX on untreated gingivitis and subgingival microbiota.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old male or female with gingivitis associated with dental plaque, no clinical signs of destructive periodontal disease, clinical attachment loss < 3mm, a minimum of 20 teeth (teeth that have gross caries, were fully crowned or extensively restored, orthodontic banded, abutments, or third molars were not included in the tooth count).

Exclusion Criteria:

* use of tobacco products, history or current manifestation of systemic disease which could impair immune response such as diabetes mellitus, immunological disorders, hepatitis and HIV infections, use of antibiotic or anti-inflammatory or immunosuppressive drugs during 3 months period prior to the start of the trial, periodontal therapy during the last 3 month, pregnancy or lactation and oral contraceptives usage.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
effectiveness of chlorhexidine mouthrinse on gingival inflammation and subgingival microbiota in addition to daily mechanical plaque control
effectiveness of chlorhexidine mouthrinse subgingival microbiota in addition to daily mechanical plaque control

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ege U School of Dentistry, Izmir, Bornova
  - Ege University School of Dentistry Dep of Periodontology, Izmir, Bornova

REFERENCES:
- [Result] Turkoglu O, Becerik S, Emingil G, Kutukculer N, Baylas H, Atilla G. The effect of adjunctive chlorhexidine mouthrinse on clinical parameters and gingival crevicular fluid cytokine levels in untreated plaque-associated gingivitis. Inflamm Res. 2009 May;58(5):277-83. doi: 10.1007/s00011-008-8129-z. PMID 19184351